CLINICAL TRIAL: NCT02386748
Title: Chewing Gums to Stimulate Intestinal Motility After Cesarean Section: A Randomized Controlled Trial
Brief Title: Chewing Gums to Stimulate Intestinal Motility After Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Collaborators: Armed Forces Hospitals, Southern Region, Saudi Arabia (Other Government)
Responsible Party: Principal Investigator, Mohamed Ellaithy, Associate professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: AFHSR 1-3-2015
Record Dates: First submitted 2015-03-05; First posted 2015-03-12 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Postoperative Care
Keywords: Cesarean section; Chewing gums; Intestinal motility
MeSH Terms: interventions — Chewing Gum; Fluid Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Chewing gum (Experimental): Chewing sugarless gum
  Interventions: Dietary Supplement: Chewing gum; Other: Intravenous fluids
- Oral fluids (Active Comparator): Clear oral fluids
  Interventions: Dietary Supplement: Oral fluids; Other: Intravenous fluids
- Intravenous fluids (Other): No chewing gum No oral fluids Only intravenous fluids (Lactated Ringer's solution)
  Interventions: Other: Intravenous fluids

INTERVENTIONS:
Dietary Supplement: Chewing gum — Chewing sugarless gum after the discharge from the operating room by two hours for at least half an hour at two hours intervals.
  Arms: Chewing gum
Dietary Supplement: Oral fluids — Starting clear oral fluids after operating room discharge by six hours, then hearing intestinal sounds on second day before initiating full regular diet.
  Arms: Oral fluids
Other: Intravenous fluids — Women in this group will not receive neither gum nor oral fluids, they will be on intravenous fluids (lactated ringer solution).

SUMMARY:
The study purpose is to evaluate the efficacy and safety of postoperative gum chewing on the recovery of intestinal movement after cesarean section.

All women undergoing elective cesarean section in King Faisal military hospital will be candidate for this trial after full explanation of the trial and informed consent to be taken from the women. Exclusion criteria will include emergency cesarean section, multifetal pregnancy, polyhydramnios, medical disorders with pregnancy, abnormal placentation (previa and/or accreta), past history of bowel injury or operation, any complications that will increase operative duration such as uterine artery injury or uterine extension.

450 consented women for being enrolled in this clinical trial and candidates for elective cesarean section will be divided into 3 groups:

* Group A, 150 women will receive sugarless gum after their operating room discharge by 2 hours for at least half an hour at two hours interval.
* Group B, 150 women will receive the traditional management of starting oral fluids after operating room discharge by 6 hours and hearing intestinal sounds on second day before initiating full regular diet.
* Group C, 150 women as control group, they will not receive neither gum nor oral fluids. They will be in intravenous fluid.

All demographic data of these women, indication of operation, operation time, type of anesthesia and pathway during hospital stay will be recovered and compared between 3 groups.

DETAILED DESCRIPTION:
Introduction; Cesarean section is the most common surgery among women which is associated with postoperative central nervous system (CNS) changes, leading to decreased bowel movements. Postoperative ileus is defined as transient cessation of coordinated bowel motility after surgical intervention. It Is one of the major problems of post-abdominal surgery which delays hospital discharge, causes abdominal pain, abdominal distension, inability to start oral feeding, breastfeeding, and eventually increases the cost of hospital care. Historically, professionals of gynecology and obstetrics waited until gut function returns allowing oral or entered feeding, characterized by symptoms such as bowel sounds, first flatus or stool, and feeling of hunger. Chewing gum can stimulate the stomach, enhances gastric secretion, increases peristaltic bowel movements and finally hastens recovery from ileus. It has also been recently considered by researchers as a strategy toward ileus reduction. It seems that a necessity is felt for more investigation on such a least-expensive physiological method in stimulating the return of bowel function.

Study purpose; To evaluate the efficacy and safety of postoperative gum chewing on the recovery of intestinal movement after cesarean section.

Intervention:

450 consented women for being enrolled in this clinical trial and candidates for elective cesarean section will be divided into 3 groups:

* Group A, 150 women will receive sugarless gum after their operating room discharge by 2 hours for at least half an hour at two hours interval.
* Group B, 150 women will receive the traditional management of starting oral fluids after operating room discharge by 6 hours and hearing intestinal sounds on second day before initiating full regular diet.
* Group C, 150 women as control group, they will not receive neither gum nor oral fluids. They will be in intravenous fluid.

All demographic data of these women, indication of operation, operation time, type of anesthesia and pathway during hospital stay will be recovered and compare between 3 groups.

Statistical Methods:

Analysis of the data will be done by IBM computer using SPSS (statistical product and service solution version 18). Quantitative variables will be described as mean with SD and median with range while Qualitative variables will be described as numbers and percentage. Chi-square test will be used to compare qualitative variables between groups. Independent sample t-test will be used to compare the groups as regard quantitative variables in parametric data (SD < 50% mean). Comparison between non-parametric groups will be done by using Mann-Whitney test. P value < 0.05 will be significant.

ELIGIBILITY:
Inclusion Criteria:

* All women undergoing elective cesarean section in King Faisal military hospital will be candidate for this trial after full explanation of the trial and informed consent to be taken from the women.

Exclusion Criteria:

* Emergency cesarean section.
* Multiple pregnancies.
* Polyhydramnios.
* Medical disorder as hypertension or diabetes mellitus.
* Abnormal placentation ,placenta previa ,accreta.
* Past history of bowel injury or operation.
* Any complications that will increase operative duration such as uterine artery injury or uterine extension.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 450 (Actual)
Dates: Start 2015-03; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Passage of stools | 72 hours

SECONDARY OUTCOMES:
Passage of flatus | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed I Ellaithy, MD, Study Chair — Armed Forces Hospital, Southern Region; Ahmed Traigey, MD, Study Director — Armed Forces Hospital, Southern Region
Locations (1):
- Postpartum ward of Armed Forces Hospital, Southern Region., Khamis Mushait, 'Asir Region, Saudi Arabia

REFERENCES:
- [Derived] Altraigey A, Ellaithy M, Atia H, Abdelrehim W, Abbas AM, Asiri M. The effect of gum chewing on the return of bowel motility after planned cesarean delivery: a randomized controlled trial. J Matern Fetal Neonatal Med. 2020 May;33(10):1670-1677. doi: 10.1080/14767058.2018.1526913. Epub 2018 Oct 29. PMID 30231787